CLINICAL TRIAL: NCT05593263
Title: Assistant Lecturer of Ophthalmology Department, Sohag University
Brief Title: Limbal Relaxing Incisions Versus Paired 4 mm Clear Corneal Incisions on Steep Meridian During Phacoemulsification
Acronym: LRI-CCI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Yasmine Gamal Abdellatife, assistant lecturer of opthalmology, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Soh-Med-22-10-17
Record Dates: First submitted 2022-10-17; First posted 2022-10-25 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Corneal Astigmatism
Keywords: astigmatism; limbal relaxing incisions; cataract surgery
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Intervention Model Description: Candidates will be randomly divided into two groups, OCCE group & LRI group before their cataract surgery.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clear corneal incisions (Experimental): the Steep meridian will be identified and marked, One clear corneal incision will be made on one side of the steep axis using 2.4mm keratome knife then enlarged to 4mm after completion of cataract surgery & other corneal 4mm incision is added to the other side of the steep axis
  Interventions: Procedure: surgical correction of astigmatism with cataract
- Limbal relaxing incision (Experimental): Single or paired LRI will be performed on the steep axis prior to phaco-emulsification procedure using a 600 μm diamond guarded blade.
  Interventions: Procedure: surgical correction of astigmatism with cataract

INTERVENTIONS:
Procedure: surgical correction of astigmatism with cataract — The Steep meridian will be identified and marked, relaxing limbal / corneal incisions will be designed according to it.

SUMMARY:
The goal of this is prospective, computer based randomized clinical trial is to compare the efficacy of reduction of the pre-existing corneal astigmatism at the time of cataract surgery in patients admitted in sohag university hospital.

the main questions it aims to answer are :

* Is limbal relaxing incisions as effective as the paired opposite 4mm clear corneal incisions technique in reduction of corneal astigmatism at the time of cataract surgery ?
* Are both techniques effective in treating mild degrees of corneal Astigmatism ?

All participants will have full ophthalmological examination necessary for routine cataract surgery, then randomly divided into 2 groups, clear corneal incision group & limbal relaxing incision group.

Researcher will compare difference between both groups regarding the following :

* Uncorrected distance visual acuity (UCVA)
* Best Corrected visual acuity (BCVA)
* keratometry readings

DETAILED DESCRIPTION:
This is prospective clinical trial will be established in Sohag university hospital. All cataract patients who will be admitted and meet the study inclusion criteria will be enrolled in this study. Candidates will be computer based randomly divided into two groups, opposite clear corneal incisions group & limbal relaxing incision group.

Inclusion criteria:

* Cataract patients aged 21- 80 years.
* keratometric astigmatism 1Diopter - 4 Diopters.
* Healthy clear cornea.

Exclusion criteria:

* History of previous keratorefractive or anterior segment surgery.
* Previous ocular trauma .
* Corneal scar or opacities.
* Irregular corneal astigmatism.
* Cataract unsuitable for phacoemulsification.
* Ongoing chronic ocular pathology

Withdrawal criteria:

* Suturing the wounds.
* Placement of more than 2 side ports.
* Any complication necessitating enlargement of the main incision.
* Wound infections.
* Second procedures within the follow-up period.
* intraocular lens tilt or in sulcus implantation.

Number of patients with adverse events, missed follow ups or changing plans will be registered and mentioned separately .

Preoperative evaluation:

Full ophthalmological examination will be done for all patients and include:

1. Uncorrected distance visual acuity (UCVA)
2. Best Corrected visual acuity (BCVA)
3. Slit lamp biomicroscopy
4. Refraction
5. Intraocular pressure measurement by (Goldman Applanation Tonometry)
6. Fundus examination.
7. keratometry (autokeratometry, Topcon KR-8900, Tokyo, Japan )
8. Pentacam (Sirius Scheimpflug Placido topography .CSO, Florence, Italy).
9. Evaluation of corneal aberrations( by IOLMaster 700 and the KR-1W Aberrometer (Topcon)

Data will be classified and saved in both hard and soft copies for secure validation and registry procedures. Two researchers will be responsible for revision of data verification to assess the accuracy of the registered data and completing it with the postoperative data.

Operative procedures:

All procedures will be performed by the same surgeon using standard phacoemulsification. All patients will have immediate pre-operative limbal-corneal marking while sitting upright and looking straight ahead using the slit lamp to avoid any cyclotorsion of the eyeball which could be induced by lying supine.

Clear corneal incisions group:

During surgery, the Steep meridian will be identified and marked using mendez ring and marker. Additional marks will be added 20 degree away from both sides of the paired incisions for further enlargement of the wound to be 4mm. One clear corneal incision will be made on one side of the steep axis using 2.4mm keratome knife (Alcon Laboratories, Inc., Fort Worth, TX ) which is kept parallel to the iris plane to maintain an incision width of approximately 1.5 mm for secure wound sealing. Routine phacoemulsification will be performed, then intraocular lens (IOL) in the bag will be inserted. Just before irrigation/aspiration (I/A) of the ophthalmic viscoelastic, a second clear corneal incision (CCI) will be made 180 degrees from the first incision. Both incisions will be extended from both sides till reaching the marking points to be exactly 4 mm by using a keratotomy knife and checked by surgical caliper.

In cases of against-the-rule (ATR) astigmatism, the opposite clear corneal incisions (OCCIs) will be made at the 3 o'clock and 9 o'clock positions. The temporal clear corneal incision will be used for phacoemulsification; the nasal CCI will not be used. In cases of with the rule astigmatism, the OCCIs will be made at the 12 o'clock and 6 o'clock positions. The superior CCI will be used for phacoemulsification; the inferior CCI will not be used. In cases of oblique astigmatism, the OCCIs will be made on the steepest meridian. The surgeon will choose the most comfortable CCI placement for phacoemulsification; the opposite symmetrical CCI will not be used. Bimanual I/A will be used in all cases. At the end of surgery, both incisions will be hydrated.

Limbal relaxing incision group:

The calculations of the length and position of LRI will be done using the Donnenfeld nomogram with the online calculator; http:// www.lricalculator.com. With the aid of pre-placed corneal reference marks (as done in the CCI group ), Single or paired LRI will be performed on the steep axis prior to phacoemulsification procedure using a 600 μm diamond guarded blade (Geuder LRI diamond knife, blade G-31468, Heidelberg, Germany ) and placed at least 0.5 mm anterior to the limbus. Using fixation ring, the eye will be fixated and the guarded knife is inserted at one end of the incision mark, as perpendicular to the corneal surface as possible, then advanced along the preset incision mark to complete the LRI trying at all times to maintain its perpendicular orientation. All patients had 2.4 mm clear corneal incision as the main phacoemulsification incision with no wound enlargement. Surgical induced astigmatism for the surgeon was previously calculated to be 0.5D which was used for the online LRI calculator.

All patients will be prescribed antibiotic and corticosteroids eye drops.

Postoperative Evaluation:

Postoperative visits will be scheduled for the first postoperative day for checking of any possible complications, then at 1 week and 1, 3, 6, months after surgery.

The data will be analysed using SPSS for Windows version 18.0 software (SPSS Inc., Chicago, IL, USA).The data will be shown as the mean and standard deviation.

Statistical analysis will be performed using the paired-samples t test to evaluate pre-operative and post-operative data within each group such as VA, keratometry reading, astigmatism and refraction. Independent-sample t test will be used to evaluate differences in astigmatism correction between OCCI and LRI groups. Vector analysis of astigmatism correction was calculated as previously described by Alpins.

ELIGIBILITY:
Inclusion Criteria:

* Cataract patients aged 21- 80 years.
* keratometric astigmatism 1D - 4D.
* Healthy clear cornea

Exclusion Criteria:

* History of previous keratorefractive or anterior segment surgery.
* Previous ocular trauma .
* Corneal scar or opacities.
* Irregular corneal astigmatism.
* Cataract unsuitable for phacoemulsification.
* Ongoing chronic ocular pathology

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-11-15 (Estimated); Primary Completion 2023-11-15 (Estimated); Study Completion 2024-02-15 (Estimated)

PRIMARY OUTCOMES:
change of corneal astigmatism assessed by K readings measurment | 1month post operative , 3 month post operative , 6 month post operative
  keratometry readings by autokeratometry, Topcon KR-8900, Tokyo, Japan ) confirmed by Pentacam (Sirius Scheimpflug Placido topography .CSO, Florence, Italy).

SECONDARY OUTCOMES:
change of manifest refraction assessed by autorefractometer (Topcon KR-8900, Tokyo, | 1month post operative , 3 month post operative , 6 month post operative
  sphere & cylinder power in diopters combined to report spherical equivalent measured by autorefractometer (Topcon KR-8900, Tokyo, Japan )